CLINICAL TRIAL: NCT07004699
Title: OPTIGO /Comparison of Two Ventilation Methods During Endoscopy of the Pharynx, Larynx and Oesophagus: Multicentre, Randomised, Non-inferiority Trial
Brief Title: Comparison of Two Ventilation Methods During Endoscopy of the Pharynx, Larynx and Oesophagus
Acronym: OPTIGO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OPTIGO
Record Dates: First submitted 2024-10-24; First posted 2025-06-04 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Oxygen Inhalation Therapy Endoscopy
MeSH Terms: interventions — Laryngoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laryngoscopy (Active Comparator)
  Interventions: Procedure: Laryngoscopy
- High-flow oxygen therapy (Experimental)
  Interventions: Procedure: High-flow oxygen therapy

INTERVENTIONS:
Procedure: Laryngoscopy — Introduction of the laryngoscope to maintain spontaneous ventilation in order to observe, in real conditions, the evolution and movements of the otorhinolaryngology sphere.
  Arms: Laryngoscopy
Procedure: High-flow oxygen therapy — Introduction of High-flow oxygen therapy to maintain spontaneous ventilation in order to observe, in real conditions, the evolution and movements of the otorhinolaryngology sphere.
  Arms: High-flow oxygen therapy

SUMMARY:
Around 15,000 ENT cancers are diagnosed each year in France. The majority of these cancers will at one time or another require an Endoscopy of the Pharynx, Larynx and Esophagus (Endo-PLE or suspension laryngoscopy). Endoscopies of the Otorhinolaryngeal (ENT) sphere are common procedures. They consist of inserting a rigid laryngoscope through the mouth, allowing full exposure of the laryngeal sphere. They are performed in most cases as part of a swelling assessment, following CT scans, or following the discovery of a mass upon palpation of the patient. Unfortunately, these are aggressive cancers that subsequently require major surgery and additional treatment by radio or chemotherapy. This examination can also be performed on patients suffering from swallowing disorders, following the appearance of polyps, and this time not requiring an adjuvant to surgery but their removal. For all patients, these endo-PLE are performed in the operating room and require general anesthesia. This surgical procedure is now performed by performing two laryngoscopies. The first is used to maintain good pulmonary oxygenation by introducing an oxygen cannula, the second constitutes the surgical procedure itself. The oxygen cannula is placed through the nasal cavity, directly up to the entrance of the vocal cords. This procedure is not without risk both for the patient (risk of dental breakage and bleeding during laryngoscopy) but also for the surgeon, because the cannula itself can obstruct his vision. It would be possible to do without one of them by setting up high-flow oxygen therapy (HFOT). This device has been widely deployed in continuous care and intensive care units, but is not yet the subject of much research in surgical units. The HFOT consists of oxygen cannulae delivering a mixture of gases at a high flow rate ranging from 20 to 70 liters per minute. The investigator want to evaluate through this study, the feasibility and effectiveness of setting up HFOT during procedures. The evaluation of this benefit compared to the standard method will be done using several elements including the collection of continuous saturation and blood analysis of capillary samples pre-, per- and post-operatively.

DETAILED DESCRIPTION:
Endoscopy involves inserting a more or less flexible camera into a natural orifice. This examination has developed considerably over the last few decades. Advances in the miniaturisation of optical elements and improvements in anaesthetic management have greatly favoured the development of this examination . It also seems important that this type of examination should be carried out on a more regular basis, in order to monitor and detect new pathologies in the population as a whole.

Cancers of all kinds are constantly on the increase. Diagnosis of these cancers has been facilitated by the development of imaging techniques, as well as by improvements in the conditions under which endoscopic examinations are carried out.

According to the French Cancer Society, ENT cancers affect an average of 15,000 new patients a year.Endoscopy of the pharynx, larynx and oesophagus (endo-PLO) is a diagnostic procedure that enables the anatomical structures that enable speech, breathing and swallowing to be visualised.

By keeping the patient on spontaneous ventilation (SV) during this procedure, the anatomical structures can be better observed. Today, this examination is carried out in operating theatres, under general anaesthetic. It is often required as part of an assessment of swelling or physiological changes in the ENT area. It is also performed in the event of a change in voice and/or the appearance of repeated discomfort when swallowing. ENT cancers are now the fourth most common type of cancer diagnosed in men. In women, there has been a marked resurgence since the increase in smoking among women, and it is expected to overtake certain digestive cancers in the coming years in terms of occurrence and diagnosis. In women, the number of ENT cancers rose by almost 157% between 1990 and 2023.

These cancers can take many forms, and affect various organs in the ENT sphere, from a bud on the vocal cords to a progressive tumour of the larynx. Endo-PLO has become an essential part of prevention and ENT surgery.

Endo-PLOs are diagnostic procedures that require a VS to be maintained. This is essential in order to be able to observe, in real conditions, the evolution and movements of the ENT sphere. The examination lasts an average of 45 minutes, from the time the patient enters the operating theatre until he or she leaves.

The patient is placed in a state of unconsciousness with loss of SV using a morphine-mimetic and a hypnotic (remifentanil and propofol) in Intravenous Targeted Anaesthesia (ITA) mode. These drugs are administered intravenously via a syringe pump, allowing narcosis to be reversed fairly quickly so that SV can be restored. Today, endo-PLO is performed using two laryngoscopies. Laryngoscopy involves inserting a curved piece of metal approximately 10 centimetres long into the patient's mouth, to expose the patient's vocal cords and insert a laryngeal device (oxygen probe, intubation probe) to enable the patient to be ventilated.

As part of an endo-PLO, an initial laryngoscopy is carried out by the State-qualified Anaesthetist Nurse or Anaesthetist Resuscitator . This first laryngoscopy is used to instil a 2% lidocaine solution (3 ml) between the vocal cords via a local anaesthetic spray device, which helps to provide intra- and post-operative analgesia. In a second stage, this first laryngoscopy will enable an oxygen cannula to be introduced via the patient's nasal cavities to the entrance to the vocal cords. Once this first laryngoscopy has been performed, the anaesthetic is gradually lifted so that the patient regains VS while remaining unconscious. A second laryngoscopy (suspension laryngoscopy) is then performed by the surgeon to proceed with the operation. Once the procedure is complete, the nasal cannula is removed and the patient awakened in the operating theatre.

In the case of ENT cancers, this tumour damage weakens the anatomical structures and encourages bleeding at the slightest contact.

As with any procedure, there is a significant risk of damage to these anatomical structures during laryngoscopy. As the tissues of the laryngeal walls are very fragile, there is a major risk of bleeding, which may cause difficulties in carrying out the surgical procedure. In addition, patients suffering from these pathologies may have other co-morbidities, requiring treatments that favour bleeding. Anti-aggregants, or blood thinners, are often prescribed for progressive cancers or heart disease. They prevent the formation of clots responsible for complications such as strokes or myocardial infarctions. On the other hand, and despite the fact that they are sometimes stopped several days before surgery, they increase the risk of bleeding during laryngoscopy.

Although this is a frequent occurrence, there are no statistics on bleeding during laryngoscopy. The fact remains, however, that this non-negligible risk adds another difficulty to the surgical procedure. In the vast majority of cases, bleeding caused by laryngoscopy is minor.

High-flow oxygen therapy (HFOT) is a medical technology that has been in use for many years, particularly at Poitiers University Hospital(6). This device enables oxygen to be administered and delivered at flow rates ranging from 20 to 70 litres per minute (L/min), with the capacity to produce an inspired fraction of oxygen (FiO2) of between 21% and 100%. It consists of a gas mixer, connected to a heater and humidifier for comfortable, optimal delivery of the gas mixture. The heater keeps the inspired gases at an average temperature of 37°C, while the humidifier prevents the patient's airways from drying out. The gas mixture comes from two different connections, linked to an air and oxygen intake, to ensure that the FiO2 recorded is the same as that delivered to the patient.

The gas mixture is propelled under pressure, via specific goggles as shown in figure 4.

OHD provides improved management of patients suffering from respiratory decompensation. It offers an alternative to non-invasive ventilation (mask ventilation) and invasive ventilation (intubation), which can sometimes be a source of anxiety and rejection for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over.
* Not requiring oxygen.
* About to undergo exclusive Endoscopy of the pharynx, larynx and oesophagus surgery.
* Score de l'American Society of Anesthesiology between 1 and 4
* Informed consent signed

Exclusion Criteria:

* Endoscopy of the pharynx, larynx and oesophagus surgery combined with another procedure
* Severe or morbid obesity (BMI ≥ 35 kg/m²)
* Patients with stage IV chronic obstructive pulmonary disease
* Allergy to one of the drugs used in anaesthesia, remifentanil and/or propofol and/or lidocaine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
The presence of oxygen desaturation ≤ 85% (Pulse Oxygen Saturation ) of the patient ≤ 85%. | up to 24 hours
  during the surgery

SECONDARY OUTCOMES:
Level of oxygenation | up to 24 hours
  Oxygenation is assessed by arterial blood gas sample
Presence of bleeding from mouth and pharynx and rupture of teeth related to laryngoscopy | up to 24 hours
  On leaving the Post Interventional Monitoring Room
Patient pain assessed | up to 24 hours
  pain is evaluated using a 100 mm visual-analogue scale, from 0, i.e "no pain", to 100 mm, i.e. "maximal imaginable pain"
The surgeon's comfort during the operation | up to 24 hours
  comfort is evaluated using a 100 mm visual-analogue scale, from 0, i.e "no discomfort", to 100 mm, i.e. "maximal imaginable discomfort"
The duration in minutes of the suspension laryngoscopy performed by the surgeon until the end of the surgical procedure | up to 24 hours
  During surgery
The duration in minutes of anaesthesia | up to 24 hours
  From induction to the patient's awakening
The cumulative dose of anaesthetics used in relation to the patient's weight | up to 24 hours
  During surgery

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume BEAUMATIN, Study Director — Poitiers University Hospital
Locations (2):
- France (2):
  - CHU Poitiers, Poitiers
  - CHU de Poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: Undecided